CLINICAL TRIAL: NCT01708746
Title: Investigation of the Impact of Noninvasive Prenatal Testing for Fetal Aneuploidy on Utilization of Prenatal Diagnostic Procedures and Pregnant Women's Views
Status: Completed | Type: Observational
Sponsor: Verinata Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VER-0008
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: High Risk Pregnancy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Enrolled subjects
- Historic control

SUMMARY:
This is a prospective, single-institution observational study to be conducted at 4 clinics within the Southern California Permanente Medical Group. Pregnant women who present for prenatal genetic counseling at the designated clinics and who meet study eligibility criteria will be offered the option of the verifi® prenatal test by a trained, licensed and certified genetic counselor (GC) . Women who elect the verifi® prenatal test will have a blood sample drawn by peripheral venipuncture that will be sent to the Verinata Health CAP-accredited clinical laboratory (Redwood City, CA). Results will be reported to the ordering health care provider by the laboratory within 8-10 business days and will be shared with the subject by their provider. Subject care and decision-making following NIPT result will be clinically managed by the provider with his/her subject and is not dictated by the study protocol. All eligible women who provide informed consent, whether they elect or decline NIPT will be asked to complete a short questionnaire on their views of prenatal testing. The uptake of invasive prenatal procedures (CVS and/or amniocentesis) by the total prospective cohort will be collected through review of electronic medical records (EMR). A historical cohort with matched demographic and pre-test indications to the prospective cohort will be identified from the EMR for comparison in the primary analysis.

ELIGIBILITY:
Inclusion Criteria

* Age 18 years or older at enrollment
* Clinically confirmed singleton pregnancy
* Gestational age between 10 weeks, 0 days and 20 weeks, 0 days
* Referred for prenatal genetic counseling due to increased risk for fetal aneuploidy (advanced maternal age (AMA ≥ 35 years at delivery, high-risk prenatal screen result, abnormal fetal ultrasound finding consistent with fetal aneuploidy, and/or history of prior affected pregnancy for fetal aneuploidy)
* Pregnancy records accessible and available for data collection (e.g., results from screening, ultrasound examinations, invasive prenatal procedures if performed, and infant hospital discharge exam)
* Able to provide consent for participation using language-appropriate forms

Exclusion Criteria

* Invasive prenatal procedure (amniocentesis or CVS) already performed
* History of demised or vanished co-twin (spontaneous or following in vitro fertilization)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is comprised of pregnant women at least 18 years of age, who meet the inclusion criteria but none of the exclusion criteria described below. Women who present for prenatal genetic counseling at one of the designated study clinics will be recruited.
Sampling Method: Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2012-11; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Invasive prenatal procedures rate measure by the occurance of chorionic villus sampling (CVS) and/or amniocentesis | Enrolled women will be evaluated on or before Gestational Age: Wk 28
  The primary objective of this study is to compare the rate of uptake of invasive prenatal procedures (chorionic villus sampling (CVS) or amniocentesis) between a prospectively enrolled cohort of pregnant women at high-risk for fetal aneuploidy who are offered noninvasive prenatal testing (NIPT; verifi® prenatal test) and a historical cohort matched for demographics and pre-test risk indications. The prospective group will include both those who accept NIPT and those who decline NIPT, but are willing to consent and complete a brief questionnaire.

SECONDARY OUTCOMES:
Preferences of pregnant women on prenatal testing by completion of preference questionnaire. | Evaluated at time of enrollment
  The secondary objective is to collect views/preferences of pregnant women on prenatal testing for fetal chromosomal abnormalities and compare results of eligible women who accept versus those who decline NIPT during the enrollment period.

CONTACTS AND LOCATIONS:
Overall Officials: George E Tiller, MD, PhD, Principal Investigator — Kaiser Permanente, Dept Genetics
Locations (4):
- United States (4):
  - Southern California Kaiser Permanente Medical Group, Baldwin Park, California
  - Southern California Kaiser Permanente Medical Group, Los Angeles, California
  - Southern California Kaiser Permanente Medical Group, Panorama City, California
  - Southern California Kaiser Permanente Medical Center, Woodland Hills, California

REFERENCES:
- [Result] Bianchi DW, Platt LD, Goldberg JD, Abuhamad AZ, Sehnert AJ, Rava RP; MatErnal BLood IS Source to Accurately diagnose fetal aneuploidy (MELISSA) Study Group. Genome-wide fetal aneuploidy detection by maternal plasma DNA sequencing. Obstet Gynecol. 2012 May;119(5):890-901. doi: 10.1097/AOG.0b013e31824fb482. PMID 22362253
- [Result] Sehnert AJ, Rhees B, Comstock D, de Feo E, Heilek G, Burke J, Rava RP. Optimal detection of fetal chromosomal abnormalities by massively parallel DNA sequencing of cell-free fetal DNA from maternal blood. Clin Chem. 2011 Jul;57(7):1042-9. doi: 10.1373/clinchem.2011.165910. Epub 2011 Apr 25. PMID 21519036